CLINICAL TRIAL: NCT01051323
Title: Non-interventional Study to Investigate Hemoglobin Levels and Dose Over Time in the Daily Use of Mircera for Renal Anemia in Larger Centers, and to Detect Differences Between Standard of Care in the Centers
Brief Title: An Observational Study of Mircera (Methoxy Polyethylene Glycol-epoetin Beta) in Patients With Renal Anemia
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22714
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Results first posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: methoxy polyethylene glycol-ep [Mircera]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-ep [Mircera] — As prescribed by physician

SUMMARY:
This observational study will investigate hemoglobin levels and Mircera (methoxy polyethyleneglycol-epoetin beta) dose over time in patients with chronic kidney disease, and compare standards of care between centers. Data from each patient will be collected over 12 months of Mircera therapy.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/= 18 years of age
* chronic kidney disease
* informed consent for data transmission

Exclusion Criteria:

* serious hematological or infectious disease
* acute bleeding in the 16 weeks preceding data collection
* participation in an interventional trial
* female patients: pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CKD patients treated with Mirecera at different medical centers
Sampling Method: Probability Sample
Enrollment: 1580 (Actual)
Dates: Start 2010-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Saarlouis, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data of this non-interventional study were analyzed by the following strata: predialysis participants versus hemodialysis participants, unless otherwise specified.
Groups:
- Methoxy Polyethylene Glycol-epoetin Beta (All Participants): Participants received methoxy polyethylene glycol-epoetin beta intravenously or subcutaneously as prescribed by the physician and were observed for 12 months. The actual dose was chosen by the physician and was adjusted as necessary.
Period: Overall Study
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (All Participants)
Started | 1580
Received at Least One Dose | 1547
Completed | 1041
Not Completed | 539
Not completed — Discontinuation of treatment | 103
Not completed — Transplantation | 28
Not completed — Dialysis dependency | 22
Not completed — Withdrawal by Subject | 13
Not completed — Lost to Follow-up | 31
Not completed — Death | 129
Not completed — Hospitalization | 28
Not completed — Other | 148
Not completed — Missing | 37

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants for whom at least one hemoglobin value after the first application of methoxy polyethylene glycol-epoetin beta during the study course was documented.
Groups:
- Methoxy Polyethylene Glycol-epoetin Beta (Predialysis): Predialysis participants received methoxy polyethylene glycol-epoetin beta intravenously or subcutaneously as prescribed by the physician and were observed for 12 months. The actual dose was chosen by the physician and was adjusted as necessary.
- Methoxy Polyethylene Glycol-epoetin Beta (Hemodialysis): Hemodialysis participants received methoxy polyethylene glycol-epoetin beta intravenously or subcutaneously as prescribed by the physician and were observed for 12 months. The actual dose was chosen by the physician and was adjusted as necessary.
- Total: Total of all reporting groups
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (Predialysis) | Methoxy Polyethylene Glycol-epoetin Beta (Hemodialysis) | Total
Number analyzed (Participants) | 326 | 1184 | 1510
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (13.3) | 68.0 (13.8) | 68.8 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 479 | 637
  Male | 168 | 705 | 873

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Hemoglobin Value Outside the Target Range
Description: Mean hemoglobin was calculated from measurements taken during the Evaluation Period (Month 0 to Month 12). The target hemoglobin range was 10 to 13 gram/deciliter (g/dL). Percentage of participants with at least one hemoglobin value less than (<) 10 g/dL or greater than (>) 13 g/dL during the evaluation period by predialysis/hemodialysis is presented.
Time Frame: Month 0 to Month 12
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (Predialysis) | Methoxy Polyethylene Glycol-epoetin Beta (Hemodialysis)
Number analyzed (Participants) | 326 | 1184
percentage of participants
  Hemoglobin value <10 g/dL | 97.9 | 72.9
  Hemoglobin value >13 g/dL | 33.7 | 35.3

2. Primary Outcome: Percentage of Participants With Hemoglobin Values Within Pre-defined Ranges During Evaluation Period by Dose Modification, Age, and Center Size
Description: The percentage of participants with hemoglobin (Hb) values within the pre-defined ranges (10-12 g/dL, 11-12 g/dL, and 11-13 g/dL) during evaluation period (Month 0 to Month 12) by dose modification (yes or no), age (<65 years, greater than or equal to [>=] 65 years) and center size (>100 participants, less than or equal to [<=] 100 participants) is presented.
Time Frame: Month 0 to Month 12
Population: FAS. n = participants evaluable for specified category for each arm group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (Predialysis) | Methoxy Polyethylene Glycol-epoetin Beta (Hemodialysis)
Number analyzed (Participants) | 326 | 1184
percentage of participants
  No dose modifications: Hb 10-12 g/dL (n=157, 242) | 11.5 | 8.7
  No dose modifications: Hb 11-12 g/dL (n=157, 242) | 0.6 | 0.8
  No dose modifications: Hb 11-13 g/dL (n=157, 242) | 11.5 | 11.2
  With dose modifications: Hb 10-12g/dL (n=169, 942) | 6.5 | 4.9
  With dose modifications: Hb 11-12g/dL (n=169, 942) | 0.6 | 0.1
  With dose modifications: Hb 11-13g/dL (n=169, 942) | 8.9 | 5.2
  Age <65 years: Hb 10-12 g/dL (n=70, 402) | 10.0 | 6.7
  Age <65 years: Hb 11-12 g/dL (n=70, 402) | 1.4 | 0.5
  Age <65 years: Hb 11-13 g/dL (n=70, 402) | 8.6 | 8.8
  Age >=65 years: Hb 10-12 g/dL (n=256, 782) | 8.6 | 5.1
  Age >=65 years: Hb 11-12 g/dL (n=256, 782) | 0.4 | 0.1
  Age >=65 years: Hb 11-13 g/dL (n=256, 782) | 10.5 | 5.4
  Center size >100: Hb 10-12 g/dL (n=99, 563) | 17.2 | 6.0
  Center size >100: Hb 11-12 g/dL (n=99, 563) | 2.0 | 0.4
  Center size >100: Hb 11-13 g/dL (n=99, 563) | 13.1 | 7.5
  Center size <=100: Hb 10-12 g/dL (n=227, 621) | 5.3 | 5.3
  Center size <=100: Hb 11-12 g/dL (n=227, 621) | 0 | 0.2
  Center size <=100: Hb 11-13 g/dL (n=227, 621) | 8.8 | 5.5

3. Primary Outcome: Percentage of Participants With Hemoglobin Values Within Pre-defined Ranges During Month 6 to Month 12 by Dose Modification, Age, and Center Size
Description: The percentage of participants with hemoglobin values within the pre-defined ranges (10-12 g/dL, 11-12 g/dL, and 11-13 g/dL) during Month 6 to Month 12 by dose modification (yes or no), age (<65 years, >=65 years) and center size (>100 participants, <=100 participants) is presented.
Time Frame: Month 6 to Month 12
Population: FAS. n = participants evaluable for specified category for each arm group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (Predialysis) | Methoxy Polyethylene Glycol-epoetin Beta (Hemodialysis)
Number analyzed (Participants) | 326 | 1184
percentage of participants
  No dose modifications: Hb 10-12 g/dL (n=157, 242) | 9.6 | 12.8
  No dose modifications: Hb 11-12 g/dL (n=157, 242) | 3.2 | 2.5
  No dose modifications: Hb 11-13 g/dL (n=157, 242) | 8.3 | 12.8
  With dose modifications: Hb 10-12g/dL (n=169, 942) | 10.7 | 14.6
  With dose modifications: Hb 11-12g/dL (n=169, 942) | 1.2 | 2.3
  With dose modifications: Hb 11-13g/dL (n=169, 942) | 9.5 | 15.1
  Age <65 years: Hb 10-12 g/dL (n=70, 402) | 11.4 | 14.7
  Age <65 years: Hb 11-12 g/dL (n=70, 402) | 4.3 | 3.0
  Age <65 years: Hb 11-13 g/dL (n=70, 402) | 12.9 | 18.4
  Age >=65 years: Hb 10-12 g/dL (n=256, 782) | 9.8 | 14.1
  Age >=65 years: Hb 11-12 g/dL (n=256, 782) | 1.6 | 2.0
  Age >=65 years: Hb 11-13 g/dL (n=256, 782) | 7.8 | 12.7
  Center size >100: Hb 10-12 g/dL (n=99, 563) | 20.2 | 14.9
  Center size >100: Hb 11-12 g/dL (n=99, 563) | 7.1 | 3.4
  Center size >100: Hb 11-13 g/dL (n=99, 563) | 15.2 | 15.1
  Center size <=100: Hb 10-12 g/dL (n=227, 621) | 5.7 | 13.7
  Center size <=100: Hb 11-12 g/dL (n=227, 621) | 0 | 1.4
  Center size <=100: Hb 11-13 g/dL (n=227, 621) | 6.2 | 14.2

4. Primary Outcome: Maximum Intra-Individual Fluctuation of Hemoglobin Values by Predialysis/Hemodialysis, Age, and Center Size
Description: For characterization of intra-individual fluctuations, the maximum absolute differences were derived from study period specific individual mean values. Maximum intra-individual fluctuation of hemoglobin values by predialysis/hemodialysis, age (<65 years, >=65 years), and center size (>100 participants, <=100 participants) is presented. Data for this outcome measure was reported for overall participants.
Time Frame: Month 0 to Month 12
Population: FAS. N (number of participants analyzed) = participants evaluable for this measure. n = participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (All Participants)
Number analyzed (Participants) | 1489
g/dL
  Predialysis (n=317) | 1.3 (0.8)
  Hemodialysis (n=1172) | 1.6 (0.8)
  Age <65 years (n=467) | 1.6 (0.8)
  Age >=65 years (n=1022) | 1.5 (0.8)
  Center size >100 participants (n=654) | 1.5 (0.8)
  Center size <=100 participants (n=835) | 1.6 (0.8)

5. Primary Outcome: Serum Ferritin Values
Description: Serum ferritin levels were measured as nanogram/milliliter (ng/mL). Data for this outcome measure was reported for overall participants.
Time Frame: Months 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
Population: FAS. N (number of participants analyzed) = participants evaluable for this measure. n = participants with serum ferritin values at each timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Methoxy Polyethylene Glycol-epoetin (All Participants): Participants received methoxy polyethylene glycol-epoetin beta intravenously or subcutaneously as prescribed by the physician and were observed for 12 months. The actual dose was chosen by the physician and was adjusted as necessary.
Arm/Group | Methoxy Polyethylene Glycol-epoetin (All Participants)
Number analyzed (Participants) | 807
ng/mL
  Month 0 (n=807) | 402.5 (365.3)
  Month 1 (n=509) | 526.5 (453.1)
  Month 2 (n=420) | 479.9 (451.5)
  Month 3 (n=399) | 412.6 (349.3)
  Month 4 (n=439) | 517.4 (423.0)
  Month 5 (n=366) | 518.2 (424.5)
  Month 6 (n=411) | 462.0 (403.9)
  Month 7 (n=443) | 567.1 (514.5)
  Month 8 (n=333) | 488.4 (414.5)
  Month 9 (n=323) | 493.0 (414.8)
  Month 10 (n=388) | 554.8 (431.0)
  Month 11 (n=307) | 542.3 (416.2)
  Month 12 (n=335) | 478.6 (354.0)

6. Primary Outcome: Serum Iron Values
Description: Serum iron levels were measured as microgram/deciliter (mcg/dL). Data for this outcome measure was reported for overall participants.
Time Frame: Months 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
Population: FAS. N (number of participants analyzed) = participants evaluable for this measure. n = participants with serum iron values at each timepoint.
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (All Participants)
Number analyzed (Participants) | 644
mcg/dL
  Month 0 (n=644) | 73.3 (65.9)
  Month 1 (n=339) | 69.5 (33.4)
  Month 2 (n=351) | 68.8 (37.1)
  Month 3 (n=375) | 74.5 (74.4)
  Month 4 (n=362) | 67.7 (31.2)
  Month 5 (n=323) | 68.9 (31.0)
  Month 6 (n=347) | 72.1 (32.7)
  Month 7 (n=362) | 74.4 (34.2)
  Month 8 (n=294) | 67.0 (31.9)
  Month 9 (n=284) | 74.3 (50.1)
  Month 10 (n=341) | 69.0 (29.2)
  Month 11 (n=263) | 64.8 (28.8)
  Month 12 (n=263) | 70.2 (29.7)

7. Primary Outcome: Transferrin Values
Description: Transferrin levels were measured as milligram/deciliter (mg/dL). Data for this outcome measure was reported for overall participants.
Time Frame: Months 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
Population: FAS. N (number of participants analyzed) = participants evaluable for this measure. n = participants with tansferrin values at each timepoint.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (All Participants)
Number analyzed (Participants) | 544
mg/dL
  Month 0 (n=544) | 196.1 (46.8)
  Month 1 (n=266) | 187.9 (40.4)
  Month 2 (n=271) | 192.5 (43.1)
  Month 3 (n=274) | 192.6 (44.2)
  Month 4 (n=292) | 187.7 (43.6)
  Month 5 (n=231) | 193.6 (41.9)
  Month 6 (n=282) | 193.9 (47.0)
  Month 7 (n=287) | 188.4 (44.0)
  Month 8 (n=199) | 192.0 (43.2)
  Month 9 (n=205) | 188.1 (44.7)
  Month 10 (n=251) | 182.3 (39.5)
  Month 11 (n=175) | 186.9 (45.1)
  Month 12 (n=179) | 189.9 (46.1)

8. Primary Outcome: Transferrin Saturation Values
Description: Transferrin saturation (TSAT) measured as a percentage, is a medical laboratory test. It is the ratio of serum iron and total iron-binding capacity, multiplied by 100. Data for this outcome measure was reported for overall participants.
Time Frame: Months 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
Population: FAS. N (number of participants analyzed) = participants evaluable for this measure. n = participants with transferrin saturation values at each timepoint.
Measure: Mean (Standard Deviation); unit: percent transferrin saturation
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (All Participants)
Number analyzed (Participants) | 489
percent transferrin saturation
  Month 0 (n=489) | 24.4 (11.8)
  Month 1 (n=298) | 27.3 (15.2)
  Month 2 (n=308) | 26.7 (13.8)
  Month 3 (n=282) | 28.0 (13.8)
  Month 4 (n=321) | 26.4 (12.9)
  Month 5 (n=276) | 27.5 (14.1)
  Month 6 (n=320) | 27.2 (13.6)
  Month 7 (n=316) | 28.2 (13.8)
  Month 8 (n=254) | 26.8 (14.0)
  Month 9 (n=241) | 27.4 (12.3)
  Month 10 (n=294) | 27.3 (12.5)
  Month 11 (n=227) | 25.7 (12.1)
  Month 12 (n=220) | 27.0 (11.8)

9. Primary Outcome: C-reactive Protein (CRP) Values
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement. Data for this outcome measure was reported for overall participants.
Time Frame: Months 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
Population: FAS. N (number of participants analyzed) = participants evaluable for this measure. n = participants with C-reactive protein values at each timepoint.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (All Participants)
Number analyzed (Participants) | 916
mg/dL
  Month 0 (n=916) | 13.3 (28.5)
  Month 1 (n=641) | 15.0 (30.7)
  Month 2 (n=529) | 12.9 (24.1)
  Month 3 (n=589) | 21.6 (119.2)
  Month 4 (n=677) | 14.5 (74.8)
  Month 5 (n=552) | 12.1 (20.6)
  Month 6 (n=567) | 15.0 (35.8)
  Month 7 (n=623) | 11.4 (19.0)
  Month 8 (n=471) | 16.5 (66.0)
  Month 9 (n=514) | 12.4 (22.0)
  Month 10 (n=535) | 11.1 (18.2)
  Month 11 (n=478) | 13.0 (29.6)
  Month 12 (n=488) | 11.2 (23.4)

10. Primary Outcome: Number of Physicians Satisfied With Treatment at Final Visit
Description: Physicians were asked to rate their satisfaction with the methoxy polyethyleneglycol-epoetin beta treatment at final visit. Physicians' responses were "very satisfied", "satisfied", "undecided", or "not satisfied". One physician could analyze multiple participants but for the purpose of analysis each physician was counted as one for each analyzed participants; hence, the number of physicians (as per this assessment) was equal to the number of participants analyzed. Data for this outcome measure was reported for overall participants.
Time Frame: Month 12 or early discontinuation
Population: FAS
Measure: Number; unit: physicians
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (All Participants)
Number analyzed (Participants) | 1510
physicians
  Very satisfied | 685
  Satisfied | 602
  Undecided | 136
  Not satisfied | 31
  Missing | 56

11. Primary Outcome: Number of Participants Who Continued Treatment With Methoxy Polyethyleneglycol-epoetin Beta After Study Completion
Description: At final visit, physicians were asked to answer ("yes" or "no") the question, whether they would continue treatment with methoxy polyethyleneglycol-epoetin beta treatment after study completion. Data for this outcome measure was reported for overall participants.
Time Frame: Month 12 or early discontinuation
Population: FAS
Measure: Number; unit: participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (All Participants)
Number analyzed (Participants) | 1510
participants
  Yes | 944
  No | 490
  Missing | 76

12. Primary Outcome: Number of Participants With Reasons for Discontinuation of Methoxy Polyethyleneglycol-epoetin Beta Treatment After Study Completion
Description: At final visit, physicians were asked to state the reasons in case of discontinuation of treatment with methoxy polyethyleneglycol-epoetin beta. The same participant could have discontinued treatment due to multiple reasons. Data for this outcome measure was reported for overall participants.
Time Frame: Month 12 or early discontinuation
Population: FAS. N (number of participants analyzed) = participants evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (All Participants)
Number analyzed (Participants) | 490
participants
  Participant's decision | 24
  Physician's decision | 177
  Insufficient efficacy | 1
  Adverse event | 5
  Missing | 10
  Death | 116
  Methoxy polyethylene glycol-epoetin not available | 57
  Organizational reasons | 34
  Hospitalization/change of medical center | 19
  Transplantation | 18
  Treatment interruption/ESA currently not necessary | 14
  High hemoglobin levels | 10
  Relocation/vacation of participant | 6
  Lost to follow-up | 6
  Dialysis | 5
  Unknown | 5
  Change of therapy | 4
  Participant does not want to continue dialysis | 1
  Therapy withdrawal | 1
  Therapy omission | 1

13. Primary Outcome: Number of Participants Who Switched to Other Erythropoiesis Stimulating Agents (ESA)-Therapy
Description: Number of participants who switched to other ESA therapies including Aranesp, Biopoin, Biosimilar, Erypo, and NeoRecormon is presented. Data for this outcome measure was reported for overall participants.
Time Frame: Month 12 or early discontinuation
Population: FAS. N (number of participants analyzed) = participants evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (All Participants)
Number analyzed (Participants) | 169
participants
  Aranesp | 30
  Biopoin | 1
  Biosimilar | 21
  Erypo | 50
  NeoRecormon | 46
  Missing | 21

14. Primary Outcome: Number of Participants Satisfied With Treatment at Final Visit
Description: Participants were asked to rate their satisfaction with methoxy polyethyleneglycol-epoetin beta treatment at final visit. Participants' responses were "very satisfied", "satisfied", "undecided", or "not satisfied". Data for this outcome measure was reported for overall participants.
Time Frame: Month 12 or early discontinuation
Population: FAS
Measure: Number; unit: participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (All Participants)
Number analyzed (Participants) | 1510
participants
  Very satisfied | 593
  Satisfied | 713
  Undecided | 114
  Not satisfied | 16
  Missing | 74

15. Secondary Outcome: Average Methoxy Polyethylene Glycol-epoetin Beta Dose
Description: Average methoxy polyethylene glycol-epoetin beta dose per application is presented by study month. Mean values were taken when more than 1 application was documented for a participant during the time period considered. Data for this outcome measure was reported for overall participants.
Time Frame: Months 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
Population: FAS. N (number of participants analyzed) = participants evaluable for this measure. n = participants with methoxy polyethylene glycol-epoetin beta dose values during each timepoint.
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (All Participants)
Number analyzed (Participants) | 1485
mcg
  Month 0 (n=1485) | 109.1 (75.9)
  Month 1 (n=1336) | 121.8 (102.2)
  Month 2 (n=1292) | 124.6 (96.7)
  Month 3 (n=1234) | 126.2 (94.1)
  Month 4 (n=1192) | 129.4 (99.8)
  Month 5 (n=1157) | 130.5 (110.2)
  Month 6 (n=1115) | 128.3 (101.7)
  Month 7 (n=1075) | 129.3 (105.1)
  Month 8 (n=1014) | 125.7 (101.9)
  Month 9 (n=993) | 122.9 (98.2)
  Month 10 (n=954) | 124.3 (101.7)
  Month 11 (n=917) | 124.5 (106.3)
  Month 12 (n=907) | 121.1 (99.1)

ADVERSE EVENTS:
Time Frame: Month 0 to Month 12
Description: Safety Analysis Set: all participants who received at least one dose of methoxy polyethylene glycol-epoetin beta during the study course.
Groups:
- Methoxy Polyethylene Glycol-epoetin Beta (Predialysis); Methoxy Polyethylene Glycol-epoetin Beta (Hemodialysis): Participants received methoxy polyethylene glycol-epoetin beta intravenously or subcutaneously as prescribed by the physician and were observed for 12 months. The actual dose was chosen by the physician and was adjusted as necessary.
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (Predialysis) | Methoxy Polyethylene Glycol-epoetin Beta (Hemodialysis)
Serious Adverse Events (participants affected / at risk) | 7/346 | 67/1201
Other Adverse Events (participants affected / at risk) | 13/346 | 196/1201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-epoetin Beta (Predialysis) (N=346) | Methoxy Polyethylene Glycol-epoetin Beta (Hemodialysis) (N=1201)
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 3
Cardiovascular disorder (Cardiac disorders) | 0 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2
Myocarditis (Cardiac disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 7
Haematemesis (Gastrointestinal disorders) | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 5
General physical health deterioration (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Ulcer haemorrhage (General disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3
Psoas abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 4
Urinary tract infection (Infections and infestations) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Haemoglobin decreased (Investigations) | 4 | 16
Platelet count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Amputation (Surgical and medical procedures) | 0 | 1
Arteriovenous shunt operation (Surgical and medical procedures) | 1 | 0
Leg amputation (Surgical and medical procedures) | 0 | 1
Nephrectomy (Surgical and medical procedures) | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-epoetin Beta (Predialysis) (N=346) | Methoxy Polyethylene Glycol-epoetin Beta (Hemodialysis) (N=1201)
Haemoglobin decreased (Investigations) | 13 | 196

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.